CLINICAL TRIAL: NCT03997201
Title: Ripple Mapping Guided Ablation of Ischaemic Ventricular Tachycardia: A Multi-centre Prospective Clinical Trial.
Brief Title: Ripple Mapping Guided Ablation of Ischaemic Ventricular Tachycardia.
Acronym: RIPPLE-VT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Barts & The London NHS Trust (Other); Papworth Hospital NHS Foundation Trust (Other Government); Nottingham University Hospitals NHS Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Hospital de Santa Maria, Portugal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18SM4892
Record Dates: First submitted 2019-06-24; First posted 2019-06-25 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Ventricular Tachycardia; Ischemic Heart Disease
Keywords: Ventricular; Tachycardia; Ischaemic; Mapping; Ablation
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Ischemia; Tachycardia; Ischemia

STUDY DESIGN:
Intervention Model Description: Prospective clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ripple Mapping guided ischaemic VT ablation (Other): Patients referred for ablation of ischaemic VT undergo Ripple Mapping guided procedure.
  Interventions: Procedure: Ripple Mapping guided ischaemic VT ablation

INTERVENTIONS:
Procedure: Ripple Mapping guided ischaemic VT ablation — Endocardial mapping of the ventricle performed with Ripple Mapping (CARTO3v6, Biosense Webster Inc). Ablation (SmarTouch Thermocool Catheter, Biosense Webster Inc) delivered to areas of abnormal "late" electrical activity within ventricular scar tissue.

SUMMARY:
The Ripple VT-1 Study is a prospective clinical trial that aims to investigate if catheter ablation of ventricular tachycardia in patients with ischaemic heart disease can be effectively performed using Ripple Mapping.

DETAILED DESCRIPTION:
Patients who have ischaemic heart disease and are at sufficient risk of, or have suffered, ventricular tachycardia may receive implantable cardioverter defibrillator (ICD) devices. ICD devices provide life-saving shocks to terminate ventricular tachycardia. There is however substantial evidence that correlates each life-saving shock with worsening prognosis.

Catheter ablation is a procedure that can treat the cause of ischaemic ventricular tachycardia (VT). Most catheter ablation procedures for ischaemic VT are performed in normal rhythm, with an end-point of arrhythmic substrate modification. Arrhythmic substrate modification refers to the process by which abnormal electrical activity in cardiac scar tissue (from ischaemic heart disease) is identified and treated by ablation.

Substrate modification catheter ablation procedures for ischaemic VT have been demonstrated to reduce ICD shocks and VT episodes in randomised trials compared to medications. However, ablation procedure outcomes are still imperfect with a recurrence rate of 50-60%.

Ripple Mapping is a method of mapping the hearts electrical signals, that may allow better identification of the abnormal activity within scar and so improve recurrence rates following ablation.

Patients referred for ablation of ischaemic VT, who have an ICD, will undergo their procedure with Ripple Mapping and subsequently followed up over a year, at 3 monthly intervals. The main assessed outcome will be ICD or VT events over a year. This will be compared to the number of ICD or VT events the year prior to ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with coronary artery disease and ischaemic cardiomyopathy requiring ICD implantation for primary or secondary prevention.
2. Any episode of VT detected or treated appropriately (within monitor zone or therapy (ATP/shock) delivered) or by 12 lead ECG if the rate below the detection level of the device. An episode of VT will be defined as lasting more than 30 secs or a regular high rate episode meeting VT criterion for >50% of the time before the first therapy is delivered (i.e. VT degenerating into VF is acceptable under these circumstances).
3. Ablation or medical therapy would be considered reasonable option for ongoing management.
4. Males or females 18 - 80 years of age.
5. Suitable candidate for catheter ablation.
6. Signed informed consent.

Exclusion Criteria:

1. Contraindication to catheter ablation.
2. VT due to reversible causes.
3. Severe valvular disease or ventricular thrombus.
4. Active gastrointestinal bleeding.
5. Serum Creatinine >200μmol/L or on dialysis.
6. Active fever or infection.
7. Life expectancy shorter than the duration of the trial.
8. Allergy to contrast.
9. Intractable heart failure (NYHA Class IV).
10. Bleeding or clotting disorders or inability to receive heparin.
11. Malignancy needing surgery, chemotherapy or radiotherapy.
12. Pregnancy or women of child-bearing potential not using a highly effective method of contraception.
13. Unable to attend follow-up visits or ICD clinics.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Combined ICD Therapies and Mortality | 12 months
  ICD therapy (ATP and shocks) for sustained ventricular tachycardia or ventricular fibrillation as documented by the patients device. Device interrogations occur 3 monthly. Combined with Mortality (all-cause) by 1 year.

SECONDARY OUTCOMES:
Achievement of the ablation procedure protocol end-point | Procedure
  Abolition of abnormal electrical activity within ischaemic ventricular scar by Ripple Mapping guided ablation
Total ICD therapy rate | 12 months
  Total appropriate and inappropriate (defined as ICD therapies for reasons other than ventricular tachycardia/fibrillation) ICD therapies (ATP and shocks).
Total VT Episodes | 12 months
  Total VT Episodes, detected by the ICD device, occurring in the 12 months after ablation
Appropriate ATP therapy rate | 12 months
  Total appropriate ICD ATP therapies during 12 month follow up after ablation
Appropriate ICD Shocks rate | 12 months
  Total ICD Shocks during 12 month follow up after ablation
Repeat catheter ablation for ischaemic ventricular tachycardia | 12 months
  Need for a repeat catheter ablation procedure after the study procedure and during the 12 month follow up period.
All cause mortality | 12 months
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Prapa Kanagaratnam, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Hammersmith Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No